CLINICAL TRIAL: NCT07292636
Title: The Effectiveness of the Twin Block and Carriere Motion Appliances in Post-pubertal Patients and an Evaluation of the Impact of Class II Malocclusion and Its Correction on Oral Health-related Quality of Life: A Randomised Controlled Trial
Brief Title: The Effectiveness of the Twin Block and Carriere Motion Appliances in Post-pubertal Patients and an Evaluation of the Impact of Class II Malocclusion and Its Correction on Oral Health-related Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aslam Alkadhimi (Other)
Collaborators: Health Service Executive, Ireland (Other); University of Dublin, Trinity College (Other); Dublin Dental University Hospital (Other)
Responsible Party: Sponsor-Investigator, Aslam Alkadhimi, PhD researcher/Consultant Orthodontist, University of Dublin, Trinity College
Organization: University of Dublin, Trinity College (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 250901
Record Dates: First submitted 2025-12-03; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: CLASS II DIVISION 1 MALOCCLUSION; Class II Malocclusion; Growth; Overjet; Class II Buccal Segment Relationship; Class II Growth Modification; Distalization; Oral Health-Related Quality of Life
Keywords: Class II Malocclusion; Overjet; Class II Molar Relationship; Class II Canine Relationship; Functional Appliance; Class II Corrector; Growth Modification; Oral Health Related Quality of Life; Twin Block; Carriere Motion Appliance; RCT
MeSH Terms: conditions — Malocclusion, Angle Class II; Overbite

STUDY DESIGN:
Intervention Model Description: Trial design: Two-arm, parallel group. Conceptual framework: Superiority trial. Allocation ration: A 1:1 allocation ratio.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of either patient or clinician will not be possible due to the nature of intervention. The trial will be single-blind, blinding will be ensured at the data collection and analysis stages in which the researchers (investigators) and statistician (outcome assessor) will be blinded to the intervention by coding all dental study casts and lateral cephalograms. The final dental study casts, lateral cephalograms and photographs will be taken (at T3) after removal of CMA and CTB so the researchers do not know which group the patients were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTB group (Active Comparator): Participants assigned to this group will receive CTB.
  Interventions: Device: CTB
- CMA group (Experimental): Participants assigned to this group will receive CMA.
  Interventions: Device: CMA

INTERVENTIONS:
Device: CTB — The appliance will be used with the bite registration taken in maximum protrusion incorporating the following features: (1) Adam's clasps on all first premolars and first permanent molars, (2) three ball-ended clasps on the mandibular incisors, (3) midline expansion screw in the maxillary component, (4) blocks intersecting at 70 degrees, with a height of 5-6 mm in the premolar region. Patients will be instructed to wear the appliance full-time, except for eating, and during contact or water sports. Objective wear time in minutes will be recorded by a Theramon® microsensor (Handelsagentur Gschladt, Hargelsberg, Austria, or Forestadent, Pforzheim, Germany) placed in the maxillary component.
  Arms: CTB group
Device: CMA — The appliance consists of rigid stainless-steel or acrylic bars bonded to the maxillary canines and first molars bilaterally. Elastics will be worn in a Class II pattern, from hooks on the maxillary canine to attachments on the mandibular first molar (bonded molar tubes). Anchorage in the mandibular dentition will be provided by an Essix-type retainer. Patients will be instructed to wear elastics full time except for eating and cleaning the teeth. The elastics protocol for the CMA appliance will be: Force 1 elastics (Henry Schein Orthodontics) that generate about 375 g of force that will be used during the first 6 weeks, changed to Force 2 elastics that generate about 540 g of force thereafter.
  Arms: CMA group

SUMMARY:
The investigators of this clinical trial aim to:

* Compare the effectiveness and efficiency of Clark's Twin Block Appliance (CTB) vs Carriere Motion Appliance (CMA) in correcting Class II malocclusion when used in post-pubertal older adolescents, in terms of skeletal and dental change.
* Evaluate potential negative oral health-related quality of life (OHRQoL) impacts during the active treatment phase with either CTB or CMA in post-pubertal adolescents.
* Investigate the impact of Class II malocclusion on oral health-related quality of life (OHRQoL) in post-pubertal adolescents.

Class II division 1 malocclusion is a dental condition where the upper teeth protrude significantly over the lower teeth. It is a common type of malocclusion observed in orthodontic practice, accounting for approximately 20-25% globally. Correcting Class II malocclusion in growing patients using functional appliances and Class II correctors is relatively predictable.

In Ireland and the United Kingdom, the Clark's Twin Block (CTB) is the most commonly used functional appliance. The CTB consists of two components: one for the upper teeth and one for the lower teeth. These components are engineered to position the lower jaw forward, thereby promoting the desired dentoskeletal changes (moving the upper teeth back and lower forward). Another device used for Class II correction is the Carriere Motion Appliance (CMA). The CMA is gaining popularity as a treatment option for Class II malocclusion, inducing dental changes similar to those achieved with a CTB. However, uncertainty persists regarding the effectiveness of these appliances in older adolescents in the post-pubertal growth phase (aged approximately 14.5 years or above).

Additionally, although both CTB and CMA are effective in growing patients in correcting dental and skeletal discrepancies, they may influence daily activities, comfort, and psychological aspects, which often results in poor compliance. Poor adherence to orthodontic treatment, whether with fixed or removable appliances, can lead to higher rates of treatment failure.

DETAILED DESCRIPTION:
Introduction:

Multiple treatment approaches are available to address the Class II byccal segment relationship characteristic of this type of malocclusion. However, the treatment approach depends on various factors, with chronological and skeletal age being pivotal. Typically, patients present with an underlying Class II skeletal pattern characterised by mandibular retrusion.

In growing patients, treatment often involves growth-dependent strategies, such as functional appliances or other Class II correctors. While these approaches primarily produce dentoalveolar effects, with less than one-third of the correction achieved by functional appliances attributable to skeletal changes, understanding the distinction between skeletal and dentoalveolar impacts is crucial. This differentiation informs treatment choice by highlighting the varying degrees to which these methods can achieve skeletal versus dental corrections, essential for tailoring patient-specific plans.

A continuing discussion exists regarding the ability of functional appliances, whether removable or fixed, to provide effective short- and long-term stimulation of mandibular growth. While this discussion endures, it is widely recognised that the majority of correction achieved with these appliances tends to be dentoalveolar rather than skeletal in nature, with only a modest proportion attributable to true mandibular advancement. Furthermore, these dentoalveolar effects are not exclusive to functional appliances, as similar outcomes have been documented with alternative Class II correctors such as the Carriere Motion Appliance, as detailed in subsequent studies.

Some researchers propose that functional appliances yield favourable outcomes by promoting mandibular growth, either through increased mandibular length or condylar growth. Conversely, other studies contend that the extent of these skeletal effects is limited. Consequently, substantial evidence indicates that dentoalveolar changes resulting from functional appliance treatment exceed the skeletal changes.

Correcting Class II malocclusion in growing patients using functional appliances and Class II correctors is relatively predictable. However, uncertainty persists regarding the effectiveness of these appliances in older adolescents in the post-pubertal growth phase (aged approximately 14.5 years or above). Limited evidence from two retrospective studies suggests that CTB and fixed functional appliances remain effective in patients with mean ages of 13.73 ± 1.51 years and 13.76 ± 1.44 years, respectively. Furthermore, a recent randomised controlled trial (RCT) demonstrated that CTB yielded comparable effects in patients aged 11 years 8 months to 12 years 8 months, relative to those who initiated treatment 18 months later. However, the interval of active treatment between the immediate treatment group and the later treatment group may not have been sufficient to reveal significant differences in treatment outcomes. The delay for the late-treatment group was constrained by the current waiting list durations in this study.

There is a notable lack of literature regarding the effectiveness of functional appliances and other Class II correctors in post-pubertal patients.

Oral Health Related Quality of Life associated with Class II and its treatment Although both CTB and CMA are effective in growing patients in correcting dental and skeletal discrepancies, they may influence daily activities, comfort, and psychological aspects, which often results in poor compliance. Poor adherence to orthodontic treatment, whether with fixed or removable appliances, can lead to higher rates of treatment failure. To address these compliance challenges, our study will use wear-time sensors in the CTBs to objectively monitor appliance adherence.

Several generic measures are used to assess oral health-related quality of life (OHRQoL) across various dental conditions. One such measure is the Child Oral Health Impact Profile (COHIP), which is also available in a short form (COHIP-19). This questionnaire is a reliable and valid tool for assessing OHRQoL in patients aged 7 to 18 years.

However, generic measures may not fully capture condition-specific impacts. To address this limitation, condition-specific OHRQoL measures have been developed. The Malocclusion Impact Questionnaire (MIQ), initially developed and tested in the UK, provides a targeted assessment of the effects of malocclusion on young patients. The Orthodontic Treatment Impact Questionnaire (OTIQ) evaluates the daily impact of orthodontic appliances on adolescents and demonstrates strong construct validity, reliability, and internal consistency.

Statement of the problem:

The effectiveness of functional appliances and Class II correctors in treating Class II malocclusion is well known. However, treating older adolescents in the post-pubertal skeletal growth phase presents certain challenges that we aim to address:

* To evaluate the effectiveness and efficiency of CTB and CMA in older adolescents who have completed their skeletal growth spurt.
* To assess the impact of CTB and CMA on OHRQoL, thereby informing treatment planning decisions and appliance wear protocols to improve treatment adherence.
* Additionally, understanding the impact of Class II malocclusion on OHRQoL may assist orthodontists in preparing patients for treatment and involving them in the decision-making process.

Importance of this research:

* The findings will provide insight into whether treatment initiated at an older age remains effective and into which of the two established treatment modalities is more effective and efficient.
* Additionally, this research will elucidate both the potential benefits on oral health-related quality of life and the challenges and adjustments young patients encounter during treatment. Such knowledge may be invaluable for orthodontists in preparing patients for treatment, refining appliance design, and improving patient comfort and adherence.
* Ultimately, these insights will inform patient selection and consent processes for older adolescent patients with Class II malocclusions.

Objectives:

The objectives of this clinical trial are to:

* Compare the amount of dental and skeletal changes and time taken to achieve those changes between post-pubertal patients wearing CTB and CMA.
* Assess the challenges and adjustments older adolescents face during CTB and CMA therapy through the completion of Orthodontic Treatment Impact Questionnaire (OTIQ).
* Evaluate the OHRQoL associated with Class II malocclusion in older adolescents through the completion of the Malocclusion Impact Questionnaire (MIQ) and the Child Oral Health Impact Profile (COHIP-19) questionnaire.

Hypotheses:

* Correction of Class II malocclusion with either CTB or CMA in post-pubertal older adolescents is effective, and both appliances are equally effective and efficient.
* Class II correction with CTB and CMA has a beneficial effect on OHRQoL in older adolescents.
* Class II malocclusion affects the OHRQoL of older adolescents negatively.

ELIGIBILITY:
Inclusion Criteria:

1. males and females aged 14 ½ -16 years from the HSE waiting list,
2. Cervical Vertebral Maturation (CVM) stage ≥5,
3. a mild-moderate skeletal II pattern,
4. normodivergent with average maxillomandibular planes angle (MMPA: 27±4 degrees),
5. Class II division 1 incisor relationship,
6. Class II molar relationship of ≥1/2 unit bilaterally,
7. overjet of ≥7 mm,
8. ≤5mm of dental crowding in both arches and
9. fluent English speaker.

Exclusion Criteria:

1. high MMPA,
2. low MMPA,
3. have/had cleft lip or palate or craniofacial syndrome,
4. hypodontia,
5. gross mandibular asymmetry,
6. a medically diagnosed growth excess or deficiency,
7. not dentally fit or
8. had previously received orthodontic treatment.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Change in molar and canine relationship at T3 (effectiveness) | T3: 9 months
  The primary outcome measure (change in molar and canine relationship) will be calculated at T3. This will be calculated by measuring the difference from T0 to T3 in the horizontal plane (in mm);
  * from the cusp tip of maxillary canine relative to the distal contact point of the opposing mandibular canine (change in canine relationship) and
  * from the mesiobuccal cusp of maxillary first molar relative to the buccal groove of mandibular first molar (change in molar relationship).
  All the measurements will be performed on dental study casts (taken at T0 and T3) articulated in maximum intercuspation position (MIP) using a vernier calliper. Measurements from right and left sides will be taken. Change in the canine and molar relationship will be calculated as the difference from T0 to T3.

SECONDARY OUTCOMES:
Change in molar and canine relationship at T2 (efficiency) | T2: 18 weeks
  The secondary outcome measure (change in molar and canine relationship) will be calculated at T2. This will be calculated by measuring the difference from T0 to T2 in the horizontal plane (in mm);
  * from the cusp tip of maxillary canine relative to the distal contact point of the opposing mandibular canine (change in canine relationship) and
  * from the mesiobuccal cusp of maxillary first molar relative to the buccal groove of mandibular first molar (change in molar relationship).
  All the measurements will be performed on intra-orally (taken at T0 and T2) using a vernier calliper. Measurements from right and left sides will be taken.
Dentoskeletal cephalometric changes at T3 | T3: 9 months
  Cephalometric dentoskeletal measurements (sagittal maxillary skeletal, sagittal mandibular skeletal, angular maxillomandibular, vertical skeletal and dentoalveolar). Each T0 and T3 lateral cephalogram will be obtained from the same machine and will be analysed by orienting it so that the Frankfurt plane is parallel to the floor, with the same magnification factor.
Impact of treatment on daily life based on the Orthodontic Treatment Impact Questionnaire (OTIQ) scores at T1 and T3 | T1: 2 weeks; T3: 9 months
  Evaluate potential negative oral health-related quality of life impacts during the active treatment phase with either CTB or CMA in post-pubertal adolescents. The Orthodontic Treatment Impact Questionnaire (OTIQ) is used to assess the day-to-day impact of any orthodontic appliance on adolescents, possessing good construct validity, reliability, and internal consistency.
  The OTIC score ranges from 0 to 44. Higher scores on the OTIQ indicate lower OHRQoL.
Impact of Class II correction on oral health-related quality of life (OHRQoL) based on the Malocclusion Impact Questionnaire (MIQ) scores at T0 and T4 | T0: Baseline; T4: 42 weeks
  The impact of Class II malocclusion on oral health-related quality of life (OHRQoL) in post-pubertal adolescents, will be investigated. The Malocclusion Impact Questionnaire (MIQ) will be used to assess this outcome.
  MIQ score ranges from 0 to 34. Higher MIQ scores indicate greater negative impact of malocclusion on OHRQoL.
Impact of Class II correction on oral health-related quality of life (OHRQoL) based on the Child Oral Health Impact Profile (COHIP-19) scores at T0 and T4 | T0: Baseline; T4: 42 weeks
  The impact of Class II malocclusion on oral health-related quality of life (OHRQoL) in post-pubertal adolescents, will be investigated. The Child Oral Health Impact Profile (COHIP), available as a short form (COHIP-19) will be used to assess this outcome.
  COHIP-19 score ranges from 0 to 76. Higher COHIP-19 score indicate greater OHRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Padhraig Fleming, Study Chair — Chair/Professor of Orthodontics. Programme Lead, Doctorate in Orthodontics. Division of Public and Child Dental Health. Dublin Dental University Hospital.; Aslam Alkadhimi, Principal Investigator — Dublin Dental Hospital, Trinity College Dublin
Locations (1):
- Ashtown Gate HSE Orthodontic Unit, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available after trial completion.
Supporting Information: Study Protocol, SAP
Time Frame: After trial completion.
Access Criteria: Journal editors upon request.